CLINICAL TRIAL: NCT01452100
Title: Efficacy of Prednisone in Patients With Severe Systemic Atheroembolism (Cholesterol Cristal Embolism)
Acronym: MECCORT
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Inclusion default
Sponsor: University Hospital, Toulouse (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1003701; 2010-021467-33 (EudraCT Number)
Record Dates: First submitted 2011-09-15; First posted 2011-10-14 (Estimated); Last update posted 2016-05-09 (Estimated); Status verified 2016-05

CONDITIONS: Cholesterol Embolism Systemic
Keywords: embolism; cholesterol cristal; creatinine; renal insufficiency; prednisone; systemic atheroembolism
MeSH Terms: conditions — Embolism; Renal Insufficiency | interventions — Prednisone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- prednisone (Experimental): • Patients enrolled into the study will be treated with prednisone, 20 mg/day (if body weight <70 kg ; or 25mg/d if body weight >70 kg) for 1 month, then tapered to 12.5 mg/d (month 2) and 7.5 mg/d (month 3) and stop. In both groups, patients will be treated according to expert advice including use of statins (according to French Health Agency recommendation), a RAS inhibitor and supportive treatment (including nutrition, treatment of heart failure, and dialysis).
  Interventions: Drug: prednisone
- placebo (Placebo Comparator): Patients enrolled into the study will be treated with placebo, 20 mg/day (if body weight <70 kg ; or 25mg/d if body weight >70 kg) for 1 month, then tapered to 12.5 mg/d (month 2) and 7.5 mg/d (month 3) and stop. In both groups, patients will be treated according to expert advice including use of statins (according to French Health Agency recommendation), a RAS inhibitor and supportive treatment (including nutrition, treatment of heart failure, and dialysis).
  Interventions: Other: placebo

INTERVENTIONS:
Drug: prednisone — Patients enrolled into the study will be treated with prednisone, 20 mg/day (if body weight <70 kg ; or 25mg/d if body weight >70 kg) for 1 month, then tapered to 12.5 mg/d (month 2) and 7.5 mg/d (month 3) and stop. In both groups, patients will be treated according to expert advice including use of statins (according to French Health Agency recommendation), a RAS inhibitor and supportive treatment (including nutrition, treatment of heart failure, and dialysis).
  Other Names: Cortancyl
  Arms: prednisone
Other: placebo — • Patients enrolled into the study will be treated with placebo, 20 mg/day (if body weight <70 kg ; or 25mg/d if body weight >70 kg) for 1 month, then tapered to 12.5 mg/d (month 2) and 7.5 mg/d (month 3) and stop. In both groups, patients will be treated according to expert advice including use of statins (according to French Health Agency recommendation), a RAS inhibitor and supportive treatment (including nutrition, treatment of heart failure, and dialysis).
  Arms: placebo

SUMMARY:
Cholesterol cristal embolization (CCE) is an orphan multisystem vascular condition occurring in elderly with severe atherosclerosis.

In most patients, avoiding the precipitating factors and combination of statin and RAS inhibitor are recommended.

The lack of randomized controlled trial in CCE precludes significant advances. The investigators decided to assess whether prednisone started early, at mild dosage and for a short period prevents death and progression to end-stage renal failure in patients with severe CCE, as compared to placebo.

DETAILED DESCRIPTION:
Erosion of atheromatous plaque results in release of cholesterol crystal embolism that ultimately occlude medium-sized arterioles and capillaries of the kidney, skin, gastrointestinal tract and central nervous system. The diagnosis relies on histopathological demonstration of cholesterol cristal embolism in any target organ, or can be assumed if the 3 following criteria are met (1) presence of one or more precipitating factors (2) renal function deterioration in atherosclerotic patients (3) ischemic changes of the extremities or demonstration of retinal CCE. Despite the dismal prognosis in multisystem CCE mortality the optimal treatment remains unknown.

In most patients, avoiding the precipitating factors and combination of statin and RAS inhibitor are recommended. The benefit of prednisone is uncertain, but its dramatic impact has been underlined in several short retrospective series, even with moderate daily dosage (0,2-0,5 mg/kg). However, adverse side effects of steroid therapy in uremic elderly with CCE have not been assessed. In addition, the optimal duration of the treatment has not been assessed. The lack of randomized controlled trial in CCE precludes significant advances. The investigators decided to assess whether prednisone started early, at mild dosage and for a short period prevents death and progression to end-stage renal failure in patients with severe CCE, as compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy-proven CCE or clinically diagnosed CCE as assessed on the 3 following criteria : presence of one or more precipitating factors renal function deterioration in atherosclerotic patients ischemic changes of the extremities or demonstration of retinal embolism
* Severe CCE as defined by either acute renal failure (S creatinine > 125 micromol/l and increase > 25 % of baseline), or severe abdominal changes (hemorrhage, infarction, perforation or weight loss > 5 % of body weight) or severe central nervous system neurological complication

Exclusion Criteria:

* CCE unproven, or restricted to one organ, or non-active contraindication to prednisone.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2011-06; Primary Completion 2015-09 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
1-year survival and 1-year renal survival (composite criteria) | 1 year

SECONDARY OUTCOMES:
Number and duration of hospitalization(s) | 1 year
  Number and duration of hospitalization(s)
course of renal function | 1 year
  stable, deterioration or improvement of serum creatinine - defined by changes > 20 % compared to base line
number of cardiovascular events | 1 year
  acute coronary syndrome, stroke, heart failure, critical lower member ischemia, digestive ischemia
prednisone tolerance | 1 year
  as regard to de novo diabetes mellitus, and severe psychiatric or infectious episode (requiring hospitalization).

CONTACTS AND LOCATIONS:
Overall Officials: Dominique Chauveau, PhD, Study Director — University Hospital, Toulouse; Antoine Huart, MPD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- CHU Toulouse service néphrologie, Toulouse, Toulouse, France

IPD SHARING:
Plan to Share IPD: No